CLINICAL TRIAL: NCT04924504
Title: Mechanisms Behind Severe Insulin Resistance During Pregnancy in Women With Glucose Metabolic Disorders (SIR-MET)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: PADME
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2; Gestational Diabetes; Overweight and Obesity; Pregnancy in Diabetic; Insulin Resistance; Insulin Sensitivity; Pregnancy, High Risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational; Overweight; Obesity; Pregnancy in Diabetics; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (maternal and umbilical) Placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type A: Healthy pregnant women without pregestational or gestational diabetes
  Interventions: Other: No interventions
- Type B: Pregnant women with type 2 diabetes or gestational diabetes with a total daily insulin dose <= 75 units/day
  Interventions: Other: No interventions
- Type C: Pregnant women with type 2 diabetes or gestational diabetes with a total daily insulin dose >= 100 units/day
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
The aim of this study is to describe the metabolic changes during pregnancy in women with type 2 diabetes or gestational diabetes in order to detect the pathophysiological mechanisms behind severe insulin resistance during pregnancy as well as the short- and long term consequences for mother and child.

Included pathophysiological mechanisms potentially associated with severe insulin resistance are: Maternal hormonal, inflammatory and metabolic markers in the blood, as well as the level, content and bioactivity of exosomes and genetic variants associated with overweight and diabetes.

In addition to the analysis on maternal blood, the same analysis will be performed on umbilical cord blood in order to determine the correlation between markers associated with insulin sensitivity in maternal and umbilical blood. Furthermore, fetal metabolic changes influence on fetal growth and development will be evaluated. Postpartum, the breast milk will also be examined for metabolic active substances that could influence the newborns growth and metabolism.

Investigating one potential short-term consequence of diabetes during pregnancy, the association between insulin resistance and structural and functional changes in the placenta will be examined as well as the consequences of such changes on fetal growth and development.

Investigating one potential long-term consequence of diabetes during pregnancy, the association between treatment with high doses of insulin during pregnancy and the future risk of developing cardiovascular diseases and heart failure will be examined.

DETAILED DESCRIPTION:
This is a prospective observational study including app. 24 pregnant women from the outpatient clinics at Department of Obstetrics and Gynecology at Aalborg and Aarhus University Hospital.

The study includes 8 healthy women without pregestational or gestational diabetes, 8 women with gestational diabetes or type 2 diabetes with a total daily insulin dose <= 75 units/day and 8 women with gestational diabetes or type 2 diabetes with a total daily insulin dose >= 100 units/day.

There are three study days: One in gestational week 28-36 (day 1), one during labour (day 2) and one 6 months postpartum (day 3).

Hormonal profiles and inflammatory markers will be measured at all three study days. During labour both maternal and umbilical blood will be collected. The blood sample analysis will include HbA1c, glukose, insulin, C-peptid, human anti-insulin antibody, lipid profile, liver enzymes, creatinine, FGF-21, TSH, Cortisol, human chorionic gonadotropin, estradiol, progesterone, SHBG, prolactin, human placental lactogen, placental growth hormone, PAPP-A, sFlt-1, PP13, IGF-1, IGF-BP's, Leptin, Adiponectin, hs-CRP, IL-6, IL-10, IL-1α, IFN-ɣ, TNF-α, ICAM1, VCAM and CD163. In addition to this, exosomes will be isolated precisely and profiling of the content of exosomes will be performed using in vitro assays. Proteomics and miRNAs sequencing will be employed. Furthermore, whole genome analysis will be applied to find genetic variants associated with overweight and diabetes (genetic analysis will not be performed on umbilical cord blood). Insulin sensitivity will be estimated using the homeostasis model assessment, IS-HOMA, based on fasting C-peptid and glucose concentrations.

In addition to the blood samples, the following examinations will be performed at day 1:

* Height, weight and bioelectrical impedance analysis
* Urine sample (Albumin-to-creatinine ratio)
* Blood pressure and 24-hour ambulatory blood pressure monitoring
* Central arterial pressure waveform analysis (SphygmoCor)
* Echocardiography
* Fetal ultrasound
* MRI scan of the placenta and heart

In addition to the blood samples, the following examinations will be performed at day 2:

* Placenta will be collected for a postpartum histopathological examination
* Breast milk (analyzed for lipid profile, leptin, adiponectin, prolactin, prolactin-binding protein, oxytocin, ghrelin, insulin, hs-CRP, IL-6, IL-10, IL-1α, IFN-ɣ, TNF-α, ICAM1, VCAM, CD163 and untargeted metabolomics)
* Skinfold measurement of the newborn with a caliper

In addition to the blood samples, the following examinations will be performed at day 3:

* Height, weight and bioelectrical impedance analysis
* Urine sample (Albumin-to-creatinine ratio)
* Blood pressure and 24-hour ambulatory blood pressure monitoring
* Central arterial pressure waveform analysis (SphygmoCor)
* Echocardiography
* Breast milk (analyzed for lipid profile, leptin, adiponectin, prolactin, prolactin-binding protein, oxytocin, ghrelin, insulin, hs-CRP, IL-6, IL-10, IL-1α, IFN-ɣ, TNF-α, ICAM1, VCAM, CD163 and untargeted metabolomics)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at The Department of Gynaecology and Obstetrics at Aarhus University Hospital or Aalborg University Hospital.
* Women have to be in 1 of 3 categories: Healthy without pregestational or gestational diabetes, type 2 diabetes treated with insulin or gestational diabetes treated with insulin.

Exclusion Criteria:

* Age < 18 years
* Not able to read and understand danish
* Previous bariatric surgery
* Treatment with systemic corticosteroids
* Other severe chronic diseases such as inflammatory bowel disease, cystic fibrosis and type 1 diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women are eligible for participation.
Study Population: The study population consist of pregnant women followed at The Department of Gynaecology and Obstetrics at Aarhus University Hospital or Aalborg University Hospital. Cases are diagnosed with gestational diabetes or pregestational type 2 diabetes and are treated with a total daily insulin dose >= 100 units/day. Controls are either healthy without pregestational or gestational diabetes or diagnosed with gestational diabetes or pregestational type 2 diabetes and are treated with a total daily insulin dose <= 75 units/day
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Association between insulin sensitivity Versus structural and functional changes in the placenta | Gestational week 28-36
  Structural and functional changes in the placenta will be evaluated using a functional T2-weighted MRI scan. Specifically the function of placenta will be evaluated using a T2-value. Furthermore, structural and functional changes in the placenta will be evaluated through a postpartum histopathological examination of the placenta. Insulin sensitivity will be estimated using the homeostasis model assessment (HOMA-IR) based on fasting C-peptid and glucose concentrations.

SECONDARY OUTCOMES:
Association between structural and functional changes in the placenta Versus fetal growth and development | Gestational week 28-36
  Structural and functional changes in the placenta will be evaluated using a functional T2-weighted MRI scan. Specifically the function of placenta will be evaluated using a T2-value. Furthermore, structural and functional changes in the placenta will be evaluated through a postpartum histopathological examination of the placenta. Fetal growth will be evaluated through a fetal ultrasound measuring biometric parameters and bloodflow.
Changes from baseline in serum or plasma concentration of metabolic, hormonal and inflammatory markers | Gestational week 28-36, at labour and 6 months postpartum
  Serum concentration of IGF-1, IGFBP-3, IGFBP-1, FGF-21, Leptin, Adiponectin, CD163, Human Chorionic Gonadotropin, Progesterone, C-peptide, Cortisol, Prolactin, Sex Hormone Binding Globulin, Estradiol, Free fatty acids, Human Placental Lactogen, Human Placental Growth Hormone, PAPP-A, sFlt-1, PP13 and human anti-insulin antibody.
  Plasma concentrations of IL-6, IL-10, IL-1alpha, IFN-gamma, TNF-alpha, ICAM1, VCAM, LDL, HDL, Triglyceride, Gamma-Glutamyl Transferase, Thyrotropin, glucose and HbA1c.
Assocation between the serum or plasma concentration of metabolic, hormonal and inflammatory markers Versus Insulin sensitivity | Gestational week 28-36, at labour and 6 months postpartum
  Association between the metabolic, hormonal and inflammatory markers listed as Outcome 2 and the Insulin sensitivity. Insulin sensitivity will be estimated using the homeostasis model assessment (HOMA-IR) based on fasting C-peptid and glucose concentrations.
Assocation between the serum or plasma concentration of metabolic, hormonal and inflammatory markers in maternal blood Versus the serum or plasma concentrations of the same markers in umbilical cord blood | At labour
  Association between the metabolic, hormonal and inflammatory markers listed as Outcome 2 in maternal and umbilical cord blood
Changes from baseline in the level, content and bioactivity of exosomes in serum and plasma. | Gestational week 28-36, at labour and 6 months postpartum
  Exosomes will be isolated and profiling of the content will be performed using SWATH mass spectrometry and miRNA sequencing.
Association between the level, content and bioactivity of exosomes in serum and plasma Versus Insulin sensitivity | Gestational week 28-36, at labour and 6 months postpartum
  Exosomes will be isolated and profiling of the content will be performed using SWATH mass spectrometry and miRNA sequencing. Insulin sensitivity will be estimated using the homeostasis model assessment (HOMA-IR) based on fasting C-peptid and glucose concentrations.
Association between the level, content and bioactivity of exosomes in serum and plasma in maternal blood Versus the level, content and bioactivity of exosomes in serum and plasma in umbilical cord blood | At labour
  Exosomes will be isolated and profiling of the content will be performed using SWATH mass spectrometry and miRNA sequencing.
Association between genetic variants related to overweight and diabetes Versus Insulin sensitivity | Gestational week 28-36
  Genetic variants will be examined using whole genome analysis (Illumina Novaseq System). Insulin sensitivity will be estimated using the homeostasis model assessment (HOMA-IR) based on fasting C-peptid and glucose concentrations.
Changes from baseline in body weight and body composition. | Gestational week 28-36 and 6 months postpartum
  Body weight measured in kilograms. Body composition: Body fat percentage and muscle mass
Changes from baseline in 24-hour ambulatory blood pressure (systolic and diastolic) | Gestational week 28-36 and 6 months postpartum
  Blood pressure includes the measurement of both systolic and diastolic blood pressure (mmHg).
Changes from baseline in cardiac function | Gestational week 28-36 and 6 months postpartum
  Cardiac function will be evaluated through an echocardiography and a MRI scan of the heart
Changes from baseline in the central aortic pressure waveform | Gestational week 28-36 and 6 months postpartum
  Central aortic pressure waveform will be evaluated through a noninvasive measurement with SphygmoCor technology

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Koefoed, MD, Principal Investigator — Aarhus University, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Aarhus N
  - Aalborg University Hospital, Aalborg

IPD SHARING:
Plan to Share IPD: No